CLINICAL TRIAL: NCT01984177
Title: Effects of Corticorelin Administration on Dopamine Transmission, Craving, and Mood in Cocaine Dependence: A [11C]-(+)-PHNO PET Investigation
Brief Title: Effects of Corticorelin Administration on Dopamine Transmission, Craving, and Mood in Cocaine Dependence
Status: Completed | Type: Observational
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Isabelle Boileau, Clinical Research Scientist, Centre for Addiction and Mental Health
Other Study IDs: 010/2012
Record Dates: First submitted 2013-10-09; First posted 2013-11-14 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Cocaine-Related Disorders; Cocaine Addiction; Substance-Related Disorders
Keywords: Cocaine; Substance-Related Disorders; Drug Addiction; Substance Addiction; Dopamine; Receptors, Dopamine D2; Receptors, Dopamine D3; Stress, Psychological; Corticorelin; Neuroendocrine System; Cortisol; Adrenocorticotropic Hormone; Positron-Emission Tomography; 11C-PHNO
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders; Stress, Psychological | interventions — Corticotropin-Releasing Hormone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- cocaine-dependent (CD): cocaine-dependent individuals
  Interventions: Drug: Corticotropin-Releasing Hormone
- healthy control (HC): healthy age and sex-matched individuals who do not use cocaine
  Interventions: Drug: Corticotropin-Releasing Hormone

INTERVENTIONS:
Drug: Corticotropin-Releasing Hormone — Each subject will receive a single dose of Corticotropin-Releasing Hormone corticorelin on a single occasion, and a volume-matched saline injection on a second occasion. Corticorelin will be administered as an intravenous infusion over a 30- to 60-second interval at a dose of 1 ug/kg body weight. ~15 minutes after Corticorelin/saline injection, [11C]-(+)-PHNO will be administered followed by 90 minutes of PET scanning. Primary outcome measure ([11C]-(+)-PHNO) as well as Secondary outcome measures (self reported feeling, hormones and physiological measures) will be obtained before saline or Corticorelin/saline injection and for 90-120 minutes following injection.
  Other Names: corticorelin

SUMMARY:
This study will, in a sample of cocaine-dependent and healthy control subjects, administer corticorelin and compare dopamine release between groups. Dopamine release will be measured using PET neuroimaging with the radiotracer [11C]-(+)-PHNO.

DETAILED DESCRIPTION:
SCIENTIFIC SUMMARY The project will, in a sample of cocaine-dependent (CD) and healthy control (HC) subjects, use administration of Corticorelin, a synthetic form of corticotropin releasing factor (CRF)and PET imaging to assess dopamine (DA) transmission in addiction. We will use [11C]-(+)-PHNO PET to measure striatal DA receptor binding on two occasions: 1) following corticorelin administration and 2) following saline. The change in receptor binding between the two occasions (i.e., displacement of [11C]-(+)-PHNO by endogenous DA) will index DA release.

SUBJECTS CD subjects will meet DSM-IV criteria for abuse or dependence and be ~10d cocaine abstinent at the time of PET. HC will be recruited to match CD on age, sex, education, and cigarette smoking.

PRIMARY OUTCOME MEASURES We will measure [11C]-(+)-PHNO binding on two occasions (corticorelin, saline), with the difference between conditions indexing dopamine release; this measure will then be compared between cocaine-dependent and control subjects. We will also measure plasma cortisol and ACTH), physiological measures, and subjective craving and mood.

ELIGIBILITY:
Inclusion Criteria:

* Sign and date informed consent
* Willing and able to complete trial as described in the protocol
* Psychiatrically healthy (as per diagnostic interview) except for cocaine dependence in cocaine users and nicotine dependence in both groups
* Mentally healthy
* Medically healthy (as per medical exam) with no current use of medications that may interfere with hormone activity or psychological measurements

Exclusion Criteria:

* Axis I psychiatric disorder (as per diagnostic interview), or medical condition that might interfere with participation in the study (as per medical exam)
* Exposure to radiation in the last 12 months exceeding the amount permissible by the CAMH PET centre
* Have received synthetic glucocorticoid or exogenous steroid therapy within one month of testing
* Exceed normal body weight
* If female: pregnancy or breast-feeding
* Metal implants or paramagnetic objects contained within the body
* Claustrophobia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: CD subjects are recruited from the local community using flyers and internet advertisements, and through referral from local clinical programs. CD subjects are recruited from the community using flyers and internet advertisements.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2013-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
PET measure: [11C]-(+)-PHNO binding | within a month following enrollment
  [11C]-(+)-PHNO binding on two occasions (following corticorelin and saline)

SECONDARY OUTCOMES:
stress hormone levels | in conjunction with PET
  plasma cortisol, ACTH
subjective measures | in conjunction with PET
  subjective stress, craving, mood, drug effects
vital signs | in conjunction with PET
  heart rate, blood pressure
neuropsychological battery | once following PET
  battery of neuropsychological tasks to assess cognitive function, general intelligence, and personality.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Boileau, PhD, Principal Investigator — Centre for Addiction and Mental Health, Research Imaging Centre
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital. It is fully affiliated with the University of Toronto, and is a PAHO/WHO Collaborating Centre — http://www.camh.ca